CLINICAL TRIAL: NCT04574154
Title: Regional Anesthesia in THR - Comparing Analgesic Efficacy of Fascia Iliaca Block and Erector Spinae Plane Block
Brief Title: Regional Anesthesia in THR - Comparing the Analgesic Efficacy of Fascia Iliaca Block and Erector Spinae Plane Block
Acronym: PTA-ALR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Dario Bugada, MD PhD, principal investigator, attending anesthesiologist, Papa Giovanni XXIII Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 191-19000
Record Dates: First submitted 2020-01-08; First posted 2020-10-05 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIB (Experimental): ultrasound guided Fascia Iliaca Block
  Interventions: Procedure: FIB; Procedure: spinal anesthesia
- ESPB (Experimental): ultrasound guided Erector Spinae Plane Block
  Interventions: Procedure: ESPB; Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: FIB — FIB with ultrasound: Ropivacaine 0.5% 40 ml
  Arms: FIB
Procedure: ESPB — ESPB (L4) with ultrasound: Ropivacaine 0.5% 40 ml
  Arms: ESPB
Procedure: spinal anesthesia — bupivacaine 0,5% 2.2 ml

SUMMARY:
THR (Total Hip Replacement) can be very painful and regional anesthesia is very effective in reducing postoperative pain. Fascia Iliaca Block (FIB) and Erector Spinae Plane Block (ESPB) are indirect approaches to the lumbar plexus that resulted to be very promising for THR. However, no studies investigated the analgesic superiority of either FIB or ESPB. In our study the investigators compare FIB and ESPB in terms of pain relief expressed as morphine consumption in the first 24 hours after primary THR.

ELIGIBILITY:
Inclusion Criteria:

* primary THR
* informed consent

Exclusion Criteria:

* allergies to study drugs
* spinal anesthesia contraindicated
* kidney failure
* epilepsy, psychiatric disease, neurologic deficits
* revision surgery
* neuropathies in the lumbar area
* no informed consent
* pregnancy
* alcohol/opioid abuse
* emergency surgery/intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
morphine | 24 hours
  milligrams of morphine consumed in the first postoperative day

SECONDARY OUTCOMES:
perceived postoperative pain: Numeric Rating Scale (NRS) | 24 hs
  11 point scale from 0 = "no pain" to 10 = "worst imaginable pain"
perceived postoperative pain: Numeric Rating Scale (NRS) | 48 hours
  11 point scale from 0 = "no pain" to 10 = "worst imaginable pain"
side effects | 48 hours
  occurrence of nausea/vomiting, ileum, pruritus and urinary retention in the first 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Aast Papa Giovanni Xxiii, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No